CLINICAL TRIAL: NCT07301229
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX43 (Anti-PD-L1 ADC) in Subjects With Advanced Pancreatic Cancer
Brief Title: A Phase II Clinical Study to Evaluate HLX43 in Subjects With Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-PDAC201
Record Dates: First submitted 2025-11-25; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX43 DOSE 1 (2.5 mg/kg) (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 1 (2.5 mg/kg)
- HLX43 DOSE 2 (3.0 mg/kg) (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 2 (3.0 mg/kg)

INTERVENTIONS:
Drug: HLX43 DOSE 1 (2.5 mg/kg) — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 1 (2.5 mg/kg)
Drug: HLX43 DOSE 2 (3.0 mg/kg) — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 DOSE 2 (3.0 mg/kg)

SUMMARY:
The study is being conducted to to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Pancreatic ductal adenocarcinoma (PDAC)

DETAILED DESCRIPTION:
This study is an open-label phase II clinical study to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Pancreatic ductal adenocarcinoma (PDAC). In this study, eligible subjects will be randomized at 1:1 ratio, and the patients will be administered with HLX43 at different doses via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study content, procedures, and potential adverse reactions before the trial, sign the informed consent form (ICF), voluntarily participate in the trial, and be able to complete the study per the protocol requirements;
2. Age ≥ 18 years, ≤75 years, at the time of signing the ICF, regardless of gender;
3. Histologically or cytologically confirmed, unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC),who has failed at least one prior line of standard systemic therapy. The prior therapy must have included a fluoropyrimidine-based or gemcitabine-based regimen;
4. At least one measurable lesion per RECIST v1.1 within 4 weeks before randomization;
5. Willing to provide archived (preferably within 2 years) or fresh tumor tissue specimens for the detection of PD-L1 expression.
6. At least 3 weeks (or 5 half-lives, whichever is shorter) since last major surgery, medical device treatment, radiotherapy (except palliative bone radiotherapy), cytotoxic chemotherapy, immunotherapy, or biological therapy; ≥2 weeks since last hormonal therapy or small molecule targeted therapy; ≥1 week since last traditional Chinese medicine treatment with anti-tumor indications or minor surgery; with treatment-related adverse events recovered to CTCAE v5.0 ≤ grade 1 (except grade 2 peripheral neuropathy and alopecia);
7. ECOG performance status 0-2 within 1 week before randomization;
8. Expected survival ≥ 3 months；
9. Adequate organ function within 1 week before randomization (no blood transfusion or colony-stimulating factors within 14 days prior to first dose)
10. Fertile participants must use ≥1 highly effective contraceptive method during the trial and for ≥6 months after last dose; females of childbearing potential must have negative pregnancy test within 7 days before enrollment.

Exclusion Criteria:

1. Histologically or cytologically confirmed as other pathological types of pancreatic cancer or containing components of other pathological differentiation;
2. Prior treatment with an antibody-drug conjugate (ADC) of topoisomerase I;
3. Received radical radiotherapy within 3 months prior to the first dose;
4. History of other malignancies within 2 years prior to randomization (except radically treated early-stage malignancies);
5. History of an adverse event that led to permanent discontinuation of prior immunotherapy, or a history of ≥ Grade 2 immune-mediated pneumonitis or immune-mediated myocarditis;
6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
7. Presence of spinal cord compression or clinically active central nervous system metastases (defined as untreated or symptomatic metastases, or those requiring corticosteroids or anticonvulsants), carcinomatous meningitis, or leptomeningeal disease;
8. History or presence of clinically significant pulmonary impairment due to concurrent lung disease, Subjects with a history of radiation pneumonitis within the past 6 months are also excluded;
9. Poorly controlled cardiovascular/cerebrovascular conditions;
10. Active systemic infections requiring IV antibiotics within 2 weeks pre-randomization;
11. Use of strong CYP2D6/CYP3A inhibitors/inducers within 2 weeks pre-randomization;
12. Systemic corticosteroid use (>10mg prednisone/day equivalent) or immunosuppressants within 2 weeks pre-randomization. Exceptions: Topical/ocular/intra-articular/nasal/inhaled steroids; short-term prophylactic use for contrast agents;
13. Active/suspected autoimmune diseases. Exceptions: Hypothyroid patients on thyroid replacement; controlled type 1 diabetes with insulin;
14. Live/attenuated vaccines within 4 weeks pre-randomization;
15. History of severe hypersensitivity to biologics/monoclonal antibodies or trial drug components;
16. Active tuberculosis;
17. Immunodeficiency disorders (HIV-positive or congenital/acquired immune deficiencies);
18. Active HBV/HCV infection or co-infection;
19. Pregnant/lactating women;
20. Undergone biliary stent placement within 7 days prior to randomization, or has unrelieved biliary or duodenal obstruction despite active treatment;
21. Suspected acute pancreatitis or a history of pancreatitis requiring clinical intervention recently;
22. Investigators' judgment of clinical/lab abnormalities or other factors making participation inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2028-02-21 (Estimated); Study Completion 2028-03-23 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks
  Objective response rate (ORR) is the proportion of subjects with the best overall response being CR or PR (assessed by investigator per RECIST v1.1)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by INV per RECIST v1.1.

SECONDARY OUTCOMES:
ORR | up to 24 week
  Objective response rate (ORR) (assessed by the IRRC per RECIST v1.1)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC per RECIST v1.1.
OS | From randomization to death from any cause (up to approximately 18 months)
  Overall Survival
DOR | up to 18 months
  Duration of response (DOR) is defined as the time from first response (CR or PR) until PD (RECIST v1.1) or death due to any cause, whichever occurs first.
DCR | up to 12 months
  Disease control rate (DCR) is defined as the proportion of subjects with a best overall response of CR, PR, or SD. Tumor response will be assessed by the investigator or IRRC as per RECIST v1.1.
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until 90 days after last dose, assessed up to 18 months
  Adverse events (AEs), serious adverse events (SAEs), laboratory tests, vital signs, 12-lead ECG, and physical examination